CLINICAL TRIAL: NCT00950612
Title: Safety and Immunogenicity Study of GSK Biologicals' Candidate Tuberculosis Vaccine (692342) When Administered to Healthy HIV-negative Adolescents Living in a TB Endemic Region
Brief Title: Safety and Immunogenicity of a Candidate Tuberculosis (TB) Vaccine in Healthy HIV Negative Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Aeras (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 112898
Record Dates: First submitted 2009-07-23; First posted 2009-08-03 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2016-11

CONDITIONS: Tuberculosis
Keywords: Tuberculosis vaccine
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Group A (Experimental)
  Interventions: Biological: GSK's investigational vaccine 692342
- Group B (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GSK's investigational vaccine 692342 — Intramuscular injection, 2 doses
  Arms: Group A
Biological: Placebo — Intramuscular injection, 2 doses
  Arms: Group B

SUMMARY:
This observer blind study will assess the safety and immunogenicity of GSK Biologicals' investigational 692342 vaccine administered at 0, 1 month to healthy adolescents living in a TB-endemic region.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and their parent(s)/ legal guardian(s) can and will comply with the requirements of the protocol.
* A male or female between, and including, 13 and 17 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject's parent(s) or legal guardian(s).
* Written informed assent obtained from the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Seronegative for HIV-1.
* No history of TB disease.
* No active pulmonary disease on chest X-ray.
* Availability for the duration of the immunisation and follow-up period, with the family not planning to move away from the study area within the next year.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject is abstinent, has practiced adequate contraception for 30 days prior to vaccination, and has a negative pregnancy test on the day of vaccination, and has agreed to continue adequate contraception during the entire vaccination period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of a registered live vaccine not foreseen by the study within 30 days preceding the first dose of study vaccine and administration of a registered inactivated vaccine within 14 days preceding the first dose of study vaccine.
* History of previous administration of investigational Mycobacterium tuberculosis vaccines.
* History of previous exposure to components of the investigational vaccine.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Any condition or illness (acute, chronic or history) or medication, which in the opinion of the investigator might interfere with the evaluation of the safety or immunogenicity of the study vaccine.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of vaccine, or planned administration during the study.
* Planned participation or participation in another experimental clinical study during the study period.
* A family history of congenital or hereditary immunodeficiency.
* Any chronic drug therapy to be continued during the study period, with the exception of vitamins and/or dietary supplements, birth control pills, anti-histamines for seasonal allergies and Specific Serotonin Reuptake Inhibitors (SSRIs).
* History of allergic reactions (significant IgE-mediated events) or anaphylaxis to any vaccine.
* History of allergic disease or reactions likely to be exacerbated by any component of the study vaccine.
* Pregnant female, lactating female or female planning to become pregnant or discontinue contraceptive precautions.
* Drug and/or alcohol abuse

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2009-12-08; Primary Completion 2010-09-30 (Actual); Study Completion 2010-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Worcester, Western Province, South Africa

REFERENCES:
- [Derived] Penn-Nicholson A, Geldenhuys H, Burny W, van der Most R, Day CL, Jongert E, Moris P, Hatherill M, Ofori-Anyinam O, Hanekom W; Vaccine Study Team; Bollaerts A, Demoitie MA, Kany Luabeya AK, De Ruymaeker E, Tameris M, Lapierre D, Scriba TJ. Safety and immunogenicity of candidate vaccine M72/AS01E in adolescents in a TB endemic setting. Vaccine. 2015 Jul 31;33(32):4025-34. doi: 10.1016/j.vaccine.2015.05.088. Epub 2015 Jun 10. PMID 26072017

RESULTS

PARTICIPANT FLOW:
Groups:
- GSK692342 Group: Healthy subjects between and including 13 to 17 years of age at the time of first vaccination, who received 2 doses of the study vaccine at Day 0 and Day 30, in the arm's deltoid region.
- Placebo Group: Healthy subjects between and including 13 to 17 years of age at the time of first vaccination, who received 2 doses of physiological saline at Day 0 and Day 30, in the arm's deltoid region.
Period: Overall Study
Arm/Group | GSK692342 Group | Placebo Group
Started | 40 | 20
Completed | 40 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK692342 Group | Placebo Group | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.8 (1.20) | 14.9 (1.12) | 14.83 (1.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 11 | 29
  Male | 22 | 9 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site. Relationship analysis was not performed.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Placebo Group
Number analyzed (Participants) | 40 | 20
Subjects
  Any Pain, Dose 1 [N=40;18] | 37 | 3
  Grade 3 Pain, Dose 1 [N=40;18] | 3 | 0
  Any Redness, Dose 1 [N=40;18] | 7 | 2
  Grade 3 Redness, Dose 1 [N=40;18] | 0 | 0
  Any Swelling, Dose 1 [N=40;18] | 14 | 2
  Grade 3 Swelling, Dose 1 [N=40;18] | 0 | 0
  Any Pain, Dose 2 [N=40;20] | 35 | 5
  Grade 3 Pain, Dose 2 [N=40;20] | 7 | 0
  Any Redness, Dose 2 [N=40;20] | 10 | 0
  Grade 3 Redness, Dose 2 [N=40;20] | 1 | 0
  Any Swelling, Dose 2 [N=40;20] | 13 | 0
  Grade 3 Swelling, Dose 2 [N=40;20] | 0 | 0
  Any Pain, Across [N=40;20] | 38 | 7
  Grade 3 Pain, Across [N=40;20] | 8 | 0
  Any Redness, Across [N=40;20] | 13 | 2
  Grade 3 Redness, Across [N=40;20] | 1 | 0
  Any Swelling, Across [N=40;20] | 20 | 2
  Grade 3 Swelling, Across [N=40;20] | 0 | 0

2. Primary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, temperature [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], gastrointestinal symptoms (gastro) [nausea, vomiting, diarrhoea and/or abdominal pain], headache, malaise and myalgia. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Placebo Group
Number analyzed (Participants) | 40 | 20
Subjects
  Any Fatigue, Dose 1 [N=40;18] | 11 | 2
  Related Fatigue, Dose 1 [N=40;18] | 11 | 2
  Grade 3 Fatigue, Dose 1 [N=40;18] | 0 | 0
  Any Gastro, Dose 1 [N=40;18] | 9 | 3
  Related Gastro, Dose 1 [N=40;18] | 9 | 3
  Grade 3 Gastro, Dose 1 [N=40;18] | 1 | 0
  Any Headache, Dose 1 [N=40;18] | 16 | 3
  Related Headache, Dose 1 [N=40;18] | 15 | 3
  Grade 3 Headache, Dose 1 [N=40;18] | 3 | 0
  Any Malaise, Dose 1 [N=40;18] | 6 | 1
  Related Malaise, Dose 1 [N=40;18] | 6 | 1
  Grade 3 Malaise, Dose 1 [N=40;18] | 0 | 0
  Any Myalgia, Dose 1 [N=40;18] | 4 | 2
  Related Myalgia, Dose 1 [N=40;18] | 4 | 2
  Grade 3 Myalgia, Dose 1 [N=40;18] | 0 | 0
  Any Temperature, Dose 1 [N=40;18] | 12 | 1
  Related Temperature, Dose 1 [N=40;18] | 11 | 1
  Grade 3 Temperature, Dose 1 [N=40;18] | 1 | 0
  Any Fatigue, Dose 2 [N=40;20] | 20 | 3
  Related Fatigue, Dose 2 [N=40;20] | 20 | 3
  Grade 3 Fatigue, Dose 2 [N=40;20] | 3 | 0
  Any Gastro, Dose 2 [N=40;20] | 13 | 2
  Related Gastro, Dose 2 [N=40;20] | 13 | 2
  Grade 3 Gastro, Dose 2 [N=40;20] | 0 | 2
  Any Headache, Dose 2 [N=40;20] | 27 | 3
  Related Headache, Dose 2 [N=40;20] | 27 | 3
  Grade 3 Headache, Dose 2 [N=40;20] | 6 | 0
  Any Malaise, Dose 2 [N=40;20] | 13 | 2
  Related Malaise, Dose 2 [N=40;20] | 13 | 2
  Grade 3 Malaise, Dose 2 [N=40;20] | 3 | 0
  Any Myalgia, Dose 2 [N=40;20] | 5 | 1
  Related Myalgia, Dose 2 [N=40;20] | 5 | 1
  Grade 3 Myalgia, Dose 2 [N=40;20] | 2 | 0
  Any Temperature, Dose 2 [N=40;20] | 24 | 1
  Related Temperature, Dose 2 [N=40;20] | 24 | 1
  Grade 3 Temperature, Dose 2 [N=40;20] | 3 | 0
  Any Fatigue, Across [N=40;20] | 21 | 5
  Related Fatigue, Across [N=40;20] | 21 | 5
  Grade 3 Fatigue, Across [N=40;20] | 3 | 0
  Any Gastro, Across [N=40;20] | 18 | 5
  Related Gastro, Across [N=40;20] | 18 | 5
  Grade 3 Gastro, Across [N=40;20] | 1 | 2
  Any Headache, Across [N=40;20] | 28 | 5
  Related Headache, Across [N=40;20] | 28 | 5
  Grade 3 Headache, Across [N=40;20] | 7 | 0
  Any Malaise, Across [N=40;20] | 14 | 3
  Related Malaise, Across [N=40;20] | 14 | 3
  Grade 3 Malaise, Across [N=40;20] | 3 | 0
  Any Myalgia, Across [N=40;20] | 7 | 2
  Related Myalgia, Across [N=40;20] | 7 | 2
  Grade 3 Myalgia, Across [N=40;20] | 2 | 0
  Any Temperature, Across [N=40;20] | 24 | 2
  Related Temperature, Across [N=40;20] | 24 | 2
  Grade 3 Temperature, Across [N=40;20] | 3 | 0

3. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset out-side the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 30-day (Days 0-29) post-vaccination period
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Placebo Group
Number analyzed (Participants) | 40 | 20
Subjects | 9 | 3

4. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 0 up to Day 210)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Placebo Group
Number analyzed (Participants) | 40 | 20
Subjects | 0 | 0

5. Primary Outcome: Number of Subjects With Normal Biochemical and Haematological Levels
Description: Among biochemical and haematological parameters assessed were alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine [CREA], haemoglobin [Hgb]. Levels of haematological/biochemical parameters assessed in terms of normal laboratory values were - normal, below and above.
Time Frame: At Day 0, 7, 30, 37 and 60
Population: The analysis was performedon the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Placebo Group
Number analyzed (Participants) | 40 | 20
Subjects
  ALT, Day 0-normal | 37 | 20
  ALT, Day 7-normal | 40 | 20
  ALT, Day 30-normal | 40 | 19
  ALT, Day 37-normal | 38 | 20
  ALT, Day 60-normal | 40 | 20
  AST, Day 0-normal | 36 | 17
  AST, Day 7-normal | 40 | 20
  AST, Day 30-normal | 38 | 20
  AST, Day 37-normal | 39 | 20
  AST, Day 60-normal | 38 | 20
  CREA, Day 0-normal | 23 | 10
  CREA, Day 7-normal | 20 | 5
  CREA, Day 30-normal | 18 | 7
  CREA, Day 37-normal | 17 | 9
  CREA, Day 60-normal | 17 | 8
  Hgb, Day 0-normal | 31 | 17
  Hgb, Day 7-normal | 28 | 16
  Hgb, Day 30-normal | 27 | 16
  Hgb, Day 37-normal | 22 | 16
  Hgb, Day 60-normal | 32 | 16

6. Primary Outcome: Number of Subjects With Normal Haematological Levels
Description: Among haematological parameters assessed were platelets [PLA], red blood cells [RBC] and white blood cells [WBC].
  Levels of haematological parameters assessed in terms of normal laboratory values were - normal, below and above.
Time Frame: At Day 0, 7, 30, 37 and 60
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Placebo Group
Number analyzed (Participants) | 40 | 20
Subjects
  PLA, Day 0-normal | 40 | 19
  PLA, Day 7-normal | 38 | 19
  PLA, Day 30-normal | 39 | 19
  PLA, Day 37-normal | 38 | 19
  PLA, Day 60-normal | 39 | 20
  RBC, Day 0-normal | 29 | 14
  RBC, Day 7-normal | 32 | 17
  RBC, Day 30-normal | 30 | 16
  RBC, Day 37-normal | 28 | 17
  RBC, Day 60-normal | 29 | 15
  WBC, Day 0-normal | 36 | 17
  WBC, Day 7-normal | 34 | 18
  WBC, Day 30-normal | 37 | 18
  WBC, Day 37-normal | 38 | 17
  WBC, Day 60-normal | 33 | 18

7. Primary Outcome: Number of Subjects With Biochemical and Haematological Above Normal Levels
Description: as for outcome 5
Time Frame: At Day 0, 7, 30, 37 and 60
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Placebo Group
Number analyzed (Participants) | 40 | 20
Subjects
  ALT, Day 0-above | 3 | 0
  ALT, Day 7- above | 0 | 0
  ALT, Day 30- above | 0 | 1
  ALT, Day 37- above | 2 | 0
  ALT, Day 60- above | 0 | 0
  AST, Day 0- above | 1 | 0
  AST, Day 7- above | 0 | 0
  AST, Day 30- above | 1 | 0
  AST, Day 37- above | 1 | 0
  AST, Day 60- above | 1 | 0
  CREA, Day 0- above | 0 | 0
  CREA, Day 7- above | 0 | 0
  CREA, Day 30- above | 0 | 0
  CREA, Day 37- above | 0 | 0
  CREA, Day 60- above | 0 | 0
  Hgb, Day 0- above | 1 | 0
  Hgb, Day 7- above | 0 | 0
  Hgb, Day 30- above | 0 | 0
  Hgb, Day 37- above | 0 | 0
  Hgb, Day 60- above | 0 | 0

8. Primary Outcome: Number of Subjects With Haematological Levels Above Normal
Description: as for outcome 6
Time Frame: At Day 0, 7, 30, 37 and 60
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Placebo Group
Number analyzed (Participants) | 40 | 20
Subjects
  PLA, Day 0-above | 0 | 1
  PLA, Day 7- above | 2 | 1
  PLA, Day 30- above | 1 | 1
  PLA, Day 37- above | 2 | 1
  PLA, Day 60- above | 1 | 0
  RBC, Day 0- above | 9 | 5
  RBC, Day 7- above | 3 | 2
  RBC, Day 30- above | 7 | 4
  RBC, Day 37- above | 7 | 2
  RBC, Day 60- above | 7 | 4
  WBC, Day 0- above | 2 | 2
  WBC, Day 7- above | 2 | 1
  WBC, Day 30- above | 0 | 2
  WBC, Day 37- above | 1 | 2
  WBC, Day 60- above | 5 | 1

9. Primary Outcome: Number of Subjects With Biochemical and Haematological Below Normal Levels
Description: as for outcome 5
Time Frame: At Day 0, 7, 30, 37 and 60
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Placebo Group
Number analyzed (Participants) | 40 | 20
Subjects
  ALT, Day 0-below | 0 | 0
  ALT, Day 7- below | 0 | 0
  ALT, Day 30-below | 0 | 0
  ALT, Day 37-below | 0 | 0
  ALT, Day 60-below | 0 | 0
  AST, Day 0-below | 0 | 0
  AST, Day 7-below | 0 | 0
  AST, Day 30-below | 0 | 0
  AST, Day 37- below | 0 | 0
  AST, Day 60- below | 0 | 0
  CREA, Day 0- below | 17 | 10
  CREA, Day 7- below | 20 | 15
  CREA, Day 30-below | 22 | 13
  CREA, Day 37-below | 23 | 11
  CREA, Day 60-below | 23 | 12
  Hgb, Day 0- below | 8 | 3
  Hgb, Day 7- below | 12 | 4
  Hgb, Day 30- below | 13 | 4
  Hgb, Day 37- below | 18 | 4
  Hgb, Day 60- below | 8 | 4

10. Primary Outcome: Number of Subjects With Haematological Levels Below Normal
Description: as for outcome 6
Time Frame: At Day 0, 7, 30, 37 and 60
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | GSK692342 Group | Placebo Group
Number analyzed (Participants) | 40 | 20
Subjects
  PLA, Day 0-below | 0 | 0
  PLA, Day 7-below | 0 | 0
  PLA, Day 30-below | 0 | 0
  PLA, Day 37-below | 0 | 0
  PLA, Day 60-below | 0 | 0
  RBC, Day 0-below | 2 | 1
  RBC, Day 7-below | 5 | 1
  RBC, Day 30-below | 3 | 0
  RBC, Day 37-below | 5 | 1
  RBC, Day 60-below | 4 | 1
  WBC, Day 0-below | 2 | 1
  WBC, Day 7-below | 4 | 1
  WBC, Day 30-below | 3 | 0
  WBC, Day 37-below | 1 | 1
  WBC, Day 60-below | 2 | 1

11. Secondary Outcome: Frequency of Mycobacterium Tuberculosis Fusion Protein (M72) Specific Cluster of Differentiation 4/8 (CD4/8+) T Cells Expressing at Least Two Different Cytokines
Description: Among cytokines expressed were interleukin-2 [IL-2], interferon-gamma [IFN-γ], tumour necrosis factor-alpha [TNF-α] and cluster of differentiation 40-ligand [CD40-L]. Analysis of cytokines expression was done by means of in vitro flow cytometry, using intracellular cytokine staining (ICS).
Time Frame: At Day 0, 7, 30, 37, 60 and 210
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects who had received at least one dose of study vaccine/placebo according to their random assignment, for whom data concerning immunogenicity outcome measures were available.
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK692342 Group | Placebo Group
Number analyzed (Participants) | 38 | 20
T cells/million cells
  CD4-All Doubles, Day 0 [N=36;17] | 200.5 [53.0 to 400.5] | 57.0 [4.0 to 402.0]
  CD4-All Doubles, Day 7 [N=32;15] | 4618.0 [554.5 to 17231.0] | 146.0 [1.0 to 352.0]
  CD4-All Doubles, Day 30 [N=38;18] | 2102.0 [946.0 to 6764.0] | 122.0 [48.0 to 227.0]
  CD4-All Doubles, Day 37 [N=37;19] | 8169.0 [4643.0 to 13735.0] | 159.0 [1.0 to 385.0]
  CD4-All Doubles, Day 60 [N=38;20] | 5621.0 [2958.0 to 8746.0] | 127.0 [32.5 to 301.5]
  CD4-All Doubles, Day 210 [N=36;20] | 2866.0 [1480.0 to 3830.0] | 113.5 [1.0 to 372.5]
  CD8-All Doubles, Day 0 [N=36;17] | 75.5 [1.0 to 173.0] | 44.0 [1.0 to 112.0]
  CD8-All Doubles, Day 7 [N=32;15] | 1515.0 [125.0 to 5802.0] | 1.0 [1.0 to 128.0]
  CD8-All Doubles, Day 30 [N=38;18] | 93.5 [1.0 to 246.0] | 15.5 [1.0 to 114.0]
  CD8-All Doubles, Day 37 [N=37;19] | 648.0 [378.0 to 1526.0] | 37.0 [1.0 to 116.0]
  CD8-All Doubles, Day 60 [N=38;20] | 113.5 [48.0 to 240.0] | 76.5 [18.0 to 111.0]
  CD8-All Doubles, Day 210 [N=36;20] | 33.5 [1.0 to 81.0] | 31.5 [1.0 to 80.0]

12. Secondary Outcome: Frequency of M72 Specific CD4+ T Cells Expressing Any Combination of Cytokines
Description: Among cytokines expressed were interleukin-2 [IL-2], interferon-gamma [IFN-γ], tumour necrosis factor-alpha [TNF-α] and cluster of differentiation 40-ligand [CD40-L], after background reduction stimulated by M72. Analysis of cytokines expression was done by means of in vitro flow cytometry, using intracellular cytokine staining (ICS).
Time Frame: At Day 0, 7, 30, 37, 60 and 210
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects who had received at least one dose of study vaccine/placebo according to their random assignment, for whom data concerning immunogenicity outcome measures were available.
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK692342 Group | Placebo Group
Number analyzed (Participants) | 39 | 20
T cells/million cells
  CD4.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(-)D0[N=38;19] | 42.0 [1.0 to 136.0] | 92.0 [1.0 to 314.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(-)D7[N=36;15] | 36.0 [1.0 to 213.0] | 1.0 [1.0 to 247.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(-)D30[N=39;20] | 172.0 [8.0 to 374.0] | 1.0 [1.0 to 77.5]
  CD4.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(-)D37[N=39;20] | 593.0 [382.0 to 944.0] | 13.5 [1.0 to 164.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(-)D60[N=38;20] | 344.0 [164.0 to 649.0] | 10.5 [1.0 to 124.5]
  CD4.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(-)D210[N=37;20] | 263.0 [112.0 to 548.0] | 46.5 [1.0 to 154.0]
  CD4.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(-)D0[N=38;19] | 1.0 [1.0 to 100.0] | 1.0 [1.0 to 21.0]
  CD4.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(-)D7[N=36;15] | 74.5 [1.0 to 236.5] | 28.0 [1.0 to 101.0]
  CD4.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(-)D30[N=39;20] | 163.0 [107.0 to 252.0] | 1.0 [1.0 to 24.0]
  CD4.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(-)D37[N=39;20] | 506.0 [306.0 to 825.0] | 17.0 [1.0 to 105.0]
  CD4.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(-)D60[N=38;20] | 296.0 [140.0 to 521.0] | 40.5 [1.0 to 72.5]
  CD4.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(-)D210[N=37;20] | 1.0 [1.0 to 107.0] | 1.0 [1.0 to 93.5]
  CD4.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(-)D0[N=38;19] | 1.0 [1.0 to 38.0] | 1.0 [1.0 to 165.0]
  CD4.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(-)D7[N=36;15] | 84.0 [1.0 to 396.0] | 20.0 [1.0 to 111.0]
  CD4.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(-)D30[N=39;20] | 1.0 [1.0 to 173.0] | 9.0 [1.0 to 114.5]
  CD4.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(-)D37[N=39;20] | 357.0 [142.0 to 648.0] | 1.0 [1.0 to 122.5]
  CD4.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(-)D60[N=38;20] | 90.5 [1.0 to 218.0] | 1.0 [1.0 to 80.0]
  CD4.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(-)D210[N=37;20] | 1.0 [1.0 to 57.0] | 1.0 [1.0 to 7.0]
  CD4.CD40L(-)+IL-2(-)+TNFα(-)+IFNγ(+)D0[N=38;19] | 68.5 [22.0 to 116.0] | 18.0 [1.0 to 165.0]
  CD4.CD40L(-)+IL-2(-)+TNFα(-)+IFNγ(+)D7[N=36;15] | 579.5 [95.0 to 1757.0] | 47.0 [1.0 to 91.0]
  CD4.CD40L(-)+IL-2(-)+TNFα(-)+IFNγ(+)D30[N=39;20] | 103.0 [27.0 to 327.0] | 32.5 [1.0 to 59.0]
  CD4.CD40L(-)+IL-2(-)+TNFα(-)+IFNγ(+)D37[N=39;20] | 871.0 [512.0 to 1624.0] | 43.0 [1.0 to 91.5]
  CD4.CD40L(-)+IL-2(-)+TNFα(-)+IFNγ(+)D60[N=38;20] | 183.5 [97.0 to 366.0] | 50.0 [22.5 to 78.5]
  CD4.CD40L(-)+IL-2(-)+TNFα(-)+IFNγ(+)D210[N=37;20] | 36.0 [1.0 to 144.0] | 1.0 [1.0 to 63.0]
  CD4.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(-)D0[N=38;19] | 1.0 [1.0 to 28.0] | 1.0 [1.0 to 24.0]
  CD4.CD40(+)+IL-2(+)+TNFα(-)+IFNγ(-)D7[N=36;15] | 95.0 [43.5 to 210.0] | 1.0 [1.0 to 48.0]
  CD4.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(-)D30[N=39;20] | 190.0 [119.0 to 350.0] | 1.0 [1.0 to 19.5]
  CD4.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(-)D37[N=39;20] | 588.0 [431.0 to 1003.0] | 11.0 [1.0 to 41.0]
  CD4.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(-)D60[N=38;20] | 375.0 [228.0 to 984.0] | 1.0 [1.0 to 27.0]
  CD4.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(-)D210[N=37;20] | 402.0 [256.0 to 920.0] | 1.0 [1.0 to 87.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(-)D0[N=38;19] | 1.0 [1.0 to 27.0] | 1.0 [1.0 to 23.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(-)D7[N=36;15] | 47.0 [1.0 to 90.5] | 1.0 [1.0 to 31.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(-)D30[N=39;20] | 23.0 [1.0 to 62.0] | 1.0 [1.0 to 1.5]
  CD4.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(-)D37[N=39;20] | 107.0 [66.0 to 169.0] | 1.0 [1.0 to 24.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(-)D60[N=38;20] | 65.5 [24.0 to 143.0] | 1.0 [1.0 to 36.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(-)D210[N=37;20] | 44.0 [13.0 to 70.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(+)D0[N=38;19] | 1.0 [1.0 to 21.0] | 1.0 [1.0 to 5.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(+)D7[N=36;15] | 120.0 [21.0 to 335.0] | 1.0 [1.0 to 34.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(+)D30[N=39;20] | 23.0 [1.0 to 48.0] | 1.0 [1.0 to 35.5]
  CD4.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(+)D37[N=39;20] | 169.0 [92.0 to 447.0] | 1.0 [1.0 to 22.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(+)D60[N=38;20] | 66.5 [21.0 to 109.0] | 1.0 [1.0 to 11.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(+)D210[N=37;20] | 70.0 [15.0 to 110.0] | 1.0 [1.0 to 14.5]

13. Secondary Outcome: Frequency of M72 Specific CD4+ T Cells Expressing Any Combination of Cytokines
Description: as for outcome 12
Time Frame: At Day 0, 7, 30, 37, 60 and 210
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK692342 Group | Placebo Group
Number analyzed (Participants) | 39 | 20
T cells/million cells
  CD4.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(-)D0[N=38;19] | 1.0 [1.0 to 31.0] | 1.0 [1.0 to 13.0]
  CD4.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(-)D7[N=36;15] | 59.0 [1.0 to 220.5] | 1.0 [1.0 to 26.0]
  CD4.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(-)D30[N=39;20] | 101.0 [18.0 to 206.0] | 1.0 [1.0 to 21.0]
  CD4.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(-)D37[N=39;20] | 248.0 [158.0 to 455.0] | 1.0 [1.0 to 24.5]
  CD4.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(-)D60[N=38;20] | 174.0 [91.0 to 377.0] | 1.0 [1.0 to 23.5]
  CD4.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(-)D210[N=37;20] | 1.0 [1.0 to 15.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(+)D0[N=38;19] | 24.5 [1.0 to 61.0] | 25.0 [1.0 to 72.0]
  CD4.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(+)D7[N=36;15] | 309.5 [64.5 to 972.0] | 29.0 [1.0 to 46.0]
  CD4.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(+)D30[N=39;20] | 66.0 [41.0 to 198.0] | 25.0 [1.0 to 44.0]
  CD4.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(+)D37[N=39;20] | 470.0 [238.0 to 874.0] | 23.5 [1.0 to 81.5]
  CD4.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(+)D60[N=38;20] | 109.0 [67.0 to 229.0] | 20.0 [1.0 to 60.0]
  CD4.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(+)D210[N=37;20] | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(+)D0[N=38;19] | 1.0 [1.0 to 28.0] | 1.0 [1.0 to 22.0]
  CD4.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(+)D7[N=36;15] | 232.5 [29.0 to 1233.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(+)D30[N=39;20] | 43.0 [1.0 to 183.0] | 1.0 [1.0 to 10.0]
  CD4.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(+)D37[N=39;20] | 314.0 [154.0 to 890.0] | 11.5 [1.0 to 45.0]
  CD4.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(+)D60[N=38;20] | 98.5 [27.0 to 258.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(+)D210[N=37;20] | 29.0 [1.0 to 113.0] | 1.0 [1.0 to 7.5]
  CD4.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(-)D0[N=38;19] | 21.0 [1.0 to 33.0] | 24.0 [1.0 to 36.0]
  CD4.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(-)D7[N=36;15] | 64.5 [20.0 to 305.5] | 1.0 [1.0 to 34.0]
  CD4.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(-)D30[N=39;20] | 131.0 [58.0 to 338.0] | 22.0 [1.0 to 49.5]
  CD4.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(-)D37[N=39;20] | 342.0 [179.0 to 549.0] | 1.0 [1.0 to 24.5]
  CD4.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(-)D60[N=38;20] | 270.0 [117.0 to 614.0] | 1.0 [1.0 to 26.5]
  CD4.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(-)D210[N=37;20] | 347.0 [157.0 to 640.0] | 21.0 [1.0 to 96.0]
  CD4.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(+)D0[N=38;19] | 1.0 [1.0 to 24.0] | 1.0 [1.0 to 27.0]
  CD4.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(+)D7[N=36;15] | 206.5 [36.0 to 692.5] | 1.0 [1.0 to 25.0]
  CD4.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(+)D30[N=39;20] | 62.0 [21.0 to 135.0] | 22.0 [1.0 to 35.5]
  CD4.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(+)D37[N=39;20] | 461.0 [133.0 to 738.0] | 1.0 [1.0 to 31.5]
  CD4.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(+)D60[N=38;20] | 118.5 [68.0 to 308.0] | 21.5 [1.0 to 42.5]
  CD4.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(+)D210[N=37;20] | 197.0 [121.0 to 340.0] | 15.5 [1.0 to 53.5]
  CD4.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(+)D0[N=38;19] | 1.0 [1.0 to 22.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(+)D7[N=36;15] | 64.5 [1.0 to 438.5] | 1.0 [1.0 to 21.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(+)D30[N=39;20] | 22.0 [1.0 to 155.0] | 1.0 [1.0 to 23.5]
  CD4.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(+)D37[N=39;20] | 112.0 [30.0 to 325.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(+)D60[N=38;20] | 59.0 [1.0 to 172.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(+)D210[N=37;20] | 45.0 [15.0 to 217.0] | 1.0 [1.0 to 17.5]
  CD4.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(+)D0[N=38;19] | 21.5 [1.0 to 86.0] | 1.0 [1.0 to 35.0]
  CD4.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(+)D7[N=36;15] | 448.5 [42.5 to 2742.5] | 1.0 [1.0 to 59.0]
  CD4.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(+)D30[N=39;20] | 97.0 [31.0 to 836.0] | 1.0 [1.0 to 56.5]
  CD4.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(+)D37[N=39;20] | 606.0 [181.0 to 1878.0] | 22.0 [1.0 to 32.5]
  CD4.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(+)D60[N=38;20] | 314.0 [111.0 to 580.0] | 22.5 [1.0 to 71.0]
  CD4.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(+)D210[N=37;20] | 15.0 [1.0 to 30.0] | 1.0 [1.0 to 1.0]
  CD4.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(+)D0[N=38;19] | 11.0 [1.0 to 46.0] | 1.0 [1.0 to 68.0]
  CD4.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(+)D7[N=36;15] | 443.0 [30.0 to 2485.5] | 21.0 [1.0 to 34.0]
  CD4.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(+)D30[N=39;20] | 121.0 [44.0 to 1202.0] | 1.0 [1.0 to 56.5]
  CD4.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(+)D37[N=39;20] | 505.0 [239.0 to 1790.0] | 43.0 [10.0 to 73.5]
  CD4.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(+)D60[N=38;20] | 346.5 [90.0 to 1102.0] | 23.5 [1.0 to 93.0]
  CD4.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(+)D210[N=37;20] | 560.0 [212.0 to 1230.0] | 49.0 [1.0 to 174.0]

14. Secondary Outcome: Frequency of M72 Specific CD8+ T Cells Expressing Any Combination of Cytokines
Description: as for outcome 12
Time Frame: At Day 0, 7, 30, 37, 60 and 210
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK692342 Group | Placebo Group
Number analyzed (Participants) | 39 | 20
T cells/million cells
  CD8.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(-)D0[N=38;19] | 20.5 [1.0 to 105.0] | 19.0 [1.0 to 182.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(-)D7[N=36;15] | 98.5 [1.0 to 186.0] | 1.0 [1.0 to 61.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(-)D30[N=39;20] | 2.0 [1.0 to 160.0] | 1.0 [1.0 to 6.5]
  CD8.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(-)D37[N=39;20] | 39.0 [1.0 to 168.0] | 42.0 [1.0 to 143.5]
  CD8.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(-)D60[N=38;20] | 5.0 [1.0 to 91.0] | 1.0 [1.0 to 141.5]
  CD8.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(-)D210[N=37;20] | 28.0 [1.0 to 92.0] | 7.0 [1.0 to 108.5]
  CD8.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(-)D0[N=38;19] | 3.5 [1.0 to 93.0] | 1.0 [1.0 to 118.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(-)D7[N=36;15] | 7.0 [1.0 to 73.5] | 1.0 [1.0 to 108.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(-)D30[N=39;20] | 26.0 [1.0 to 106.0] | 5.5 [1.0 to 60.5]
  CD8.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(-)D37[N=39;20] | 13.0 [1.0 to 94.0] | 35.5 [1.0 to 118.5]
  CD8.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(-)D60[N=38;20] | 40.0 [1.0 to 131.0] | 109.5 [1.0 to 142.5]
  CD8.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(-)D210[N=37;20] | 4.0 [1.0 to 107.0] | 34.5 [1.0 to 101.5]
  CD8.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(-)D0[N=38;19] | 16.5 [1.0 to 71.0] | 1.0 [1.0 to 66.0]
  CD8.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(-)D7[N=36;15] | 1.0 [1.0 to 94.0] | 8.0 [1.0 to 130.0]
  CD8.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(-)D30[N=39;20] | 1.0 [1.0 to 62.0] | 1.0 [1.0 to 47.5]
  CD8.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(-)D37[N=39;20] | 1.0 [1.0 to 46.0] | 1.0 [1.0 to 50.0]
  CD8.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(-)D60[N=38;20] | 1.0 [1.0 to 74.0] | 8.0 [1.0 to 40.5]
  CD8.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(-)D210[N=37;20] | 1.0 [1.0 to 36.0] | 1.0 [1.0 to 43.0]
  CD8.CD40L(-)+IL-2(-)+TNFα(-)+IFNγ(+)D0[N=38;19] | 66.0 [1.0 to 182.0] | 87.0 [1.0 to 196.0]
  CD8.CD40L(-)+IL-2(-)+TNFα(-)+IFNγ(+)D7[N=36;15] | 303.0 [84.0 to 541.0] | 109.0 [1.0 to 186.0]
  CD8.CD40L(-)+IL-2(-)+TNFα(-)+IFNγ(+)D30[N=39;20] | 93.0 [1.0 to 143.0] | 76.5 [26.0 to 256.0]
  CD8.CD40L(-)+IL-2(-)+TNFα(-)+IFNγ(+)D37[N=39;20] | 190.0 [33.0 to 301.0] | 95.0 [7.0 to 321.5]
  CD8.CD40L(-)+IL-2(-)+TNFα(-)+IFNγ(+)D60[N=38;20] | 70.5 [21.0 to 261.0] | 104.5 [32.5 to 296.0]
  CD8.CD40L(-)+IL-2(-)+TNFα(-)+IFNγ(+)D210[N=37;20] | 61.0 [1.0 to 135.0] | 37.5 [1.0 to 104.5]
  CD8.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(-)D0[N=38;19] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(-)D7[N=36;15] | 1.0 [1.0 to 33.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(-)D30[N=39;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(-)D37[N=39;20] | 1.0 [1.0 to 46.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(-)D60[N=38;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(-)D210[N=37;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(-)D0[N=38;19] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(-)D7[N=36;15] | 1.0 [1.0 to 10.5] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(-)D30[N=39;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(-)D37[N=39;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(-)D60[N=38;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(-)D210[N=37;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(+)D0[N=38;19] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 27.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(+)D7[N=36;15] | 94.0 [1.0 to 257.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(+)D30[N=39;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(+)D37[N=39;20] | 33.0 [1.0 to 187.0] | 1.0 [1.0 to 10.5]
  CD8.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(+)D60[N=38;20] | 1.0 [1.0 to 28.0] | 1.0 [1.0 to 39.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(-)+IFNγ(+)D210[N=37;20] | 24.0 [1.0 to 51.0] | 18.5 [1.0 to 74.5]

15. Secondary Outcome: Frequency of M72 Specific CD8+ T Cells Expressing Any Combination of Cytokines
Description: as for outcome 12
Time Frame: At Day 0, 7, 30, 37, 60 and 210
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | GSK692342 Group | Placebo Group
Number analyzed (Participants) | 39 | 20
T cells/million cells
  CD8.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(-)D0[N=38;19] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(-)D7[N=36;15] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(-)D30[N=39;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(-)D37[N=39;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 9.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(-)D60[N=38;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(-)D210[N=37;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(+)D0[N=38;19] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(+)D7[N=36;15] | 1.0 [1.0 to 30.0] | 1.0 [1.0 to 18.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(+)D30[N=39;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(+)D37[N=39;20] | 1.0 [1.0 to 37.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(+)D60[N=38;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(-)+IFNγ(+)D210[N=37;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(+)D0[N=38;19] | 1.0 [1.0 to 36.0] | 1.0 [1.0 to 25.0]
  CD8.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(+)D7[N=36;15] | 78.5 [1.0 to 244.5] | 1.0 [1.0 to 26.0]
  CD8.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(+)D30[N=39;20] | 1.0 [1.0 to 51.0] | 1.0 [1.0 to 28.0]
  CD8.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(+)D37[N=39;20] | 36.0 [1.0 to 79.0] | 10.5 [1.0 to 73.0]
  CD8.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(+)D60[N=38;20] | 21.0 [1.0 to 65.0] | 1.0 [1.0 to 24.5]
  CD8.CD40L(-)+IL-2(-)+TNFα(+)+IFNγ(+)D210[N=37;20] | 1.0 [1.0 to 20.0] | 1.0 [1.0 to 6.5]
  CD8.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(-)D0[N=38;19] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(-)D7[N=36;15] | 1.0 [1.0 to 27.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(-)D30[N=39;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(-)D37[N=39;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(-)D60[N=38;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(-)D210[N=37;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(+)D0[N=38;19] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(+)D7[N=36;15] | 41.5 [1.0 to 170.5] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(+)D30[N=39;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(+)D37[N=39;20] | 22.0 [1.0 to 66.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(+)D60[N=38;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(-)+IFNγ(+)D210[N=37;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(+)D0[N=38;19] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(+)D7[N=36;15] | 105.5 [1.0 to 435.5] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(+)D30[N=39;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(+)D37[N=39;20] | 22.0 [1.0 to 96.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(+)D60[N=38;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(-)+TNFα(+)+IFNγ(+)D210[N=37;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(+)D0[N=38;19] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(+)D7[N=36;15] | 51.0 [1.0 to 129.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(+)D30[N=39;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(+)D37[N=39;20] | 1.0 [1.0 to 38.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(+)D60[N=38;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(-)+IL-2(+)+TNFα(+)+IFNγ(+)D210[N=37;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(+)D0[N=38;19] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(+)D7[N=36;15] | 184.0 [1.0 to 577.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(+)D30[N=39;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(+)D37[N=39;20] | 37.0 [1.0 to 140.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(+)D60[N=38;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  CD8.CD40L(+)+IL-2(+)+TNFα(+)+IFNγ(+)D210[N=37;20] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

16. Secondary Outcome: Anti-M72 Specific Antibody Concentrations
Description: Antibody concentrations given in Enzyme-Linked Immunosorbent Assay (ELISA) units per millilitre (EL.U/mL) were expressed as Geometric Mean Concentrations (GMCs).
Time Frame: At Day 0, 30, 60 and 210
Population: as for outcome 12
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK692342 Group | Placebo Group
Number analyzed (Participants) | 39 | 20
EL.U/mL
  Anti-M72, D0 | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4]
  Anti-M72, D30 | 22.2 [15.3 to 32.4] | 1.6 [1.2 to 2.2]
  Anti-M72, D60 | 1077.8 [828.3 to 1402.5] | 1.8 [1.3 to 2.4]
  Anti-M72, D210 | 121.9 [93.5 to 159.1] | 1.5 [1.3 to 1.7]

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms during the 7-day post vaccination period (Days 0-6); AEs during the 30-day post vaccination period (Days 0-29), SAEs up to Day 210
Arm/Group | GSK692342 Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/20
Other Adverse Events (participants affected / at risk) | 38/40 | 15/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK692342 Group (N=40) | Placebo Group (N=20)
Pain (General disorders) | 38 | 7
Redness (millimeters) (General disorders) | 13 | 2
Swelling (millimeters) (General disorders) | 20 | 2
Fatigue (General disorders) | 21 | 5
Gastrointestinal (General disorders) | 18 | 5
Headache (General disorders) | 28 | 5
Malaise (General disorders) | 14 | 3
Myalgia (General disorders) | 7 | 2
Temperature/(Orally) (°C) (General disorders) | 24 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Haemoglobin decreased (Investigations) | 2 | 0
White blood cell count decreased (Investigations) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.